CLINICAL TRIAL: NCT02040350
Title: Study Effect of WHO Recommended Dose of Pralidoxime in the Treatment of Organophosphorus Poisoning
Brief Title: Is the WHO Recommended Dose of Pralidoxime Effective in the Treatment of Organophosphorus Poisoning?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tariq Wani, Registar, Sheri Kashmir Institute of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1151-9883
Record Dates: First submitted 2014-01-09; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Deaths
Keywords: Pralidoxime, atropine, organophosphorous poisoning.
MeSH Terms: conditions — Death | interventions — pralidoxime; Oximes

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo was given to compare the effects
  Interventions: Drug: Pralidoxime
- Pralidoxime (Active Comparator): Pralidoxime for treating organophosphorous poisoning patients
  Interventions: Drug: Pralidoxime

INTERVENTIONS:
Drug: Pralidoxime — Pralidoxime was compared to placebo to study the effects of the drug on mortatlity
  Other Names: Oximes

SUMMARY:
To evaluate the effectiveness of Pralidoxime, a drug used for treatment of pesticide poisoning (Organophosphorous poisonings)

DETAILED DESCRIPTION:
The present study was designed to critically analyze the role of pralidoxime in patients with moderate to severe poisoning by dividing them into two comparable groups in all aspects and using WHO recommended dose of pralidoxime (30mg/kg bolus I.V over 20 min followed by 8mg/kg/hr continuous infusion). This dose and continuous infusion protocol is more likely to maintain adequate blood concentrations of pralidoxime throughout 24 hours and thus would avoid any failures in effectiveness of pralidoxime because of inconsistent blood levels.

ELIGIBILITY:
Inclusion Criteria:

history of alleged organophosphorus intake age > 14 years < 60 years clinical signs and symptoms of organophosphorus poisoning.

Exclusion Criteria:

< 14 years or > 60 years of age known pregnancy pralidoxime administration at the transferring hospital carbamate poisoning any chronic illnesses

≥ 12 hour interval from time of poisoning to initiation of treatment pre-hospital cardiac or respiratory arrest.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
mortality rate | upto one year

SECONDARY OUTCOMES:
duration of ventilation | upto one year

OTHER OUTCOMES:
duration of ICU stay | upto one year

CONTACTS AND LOCATIONS:
Overall Officials: Showkat Gurcoo, MD, Study Director — SKIMS
Locations (1):
- Sheri kashmir insititute of medical sciences, Srinagar, Srinagar Kashmir, India

REFERENCES:
- [Background] Eddleston M, Buckley NA, Eyer P, Dawson AH. Management of acute organophosphorus pesticide poisoning. Lancet. 2008 Feb 16;371(9612):597-607. doi: 10.1016/S0140-6736(07)61202-1. PMID 17706760